CLINICAL TRIAL: NCT06910267
Title: Leveraging Adult Protective Service Interaction to Offer Evidence-Based Treatment for Depression in Elder Neglect/Self Neglect
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Leila Wood, professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-24-1021; 1P30AG086563-01 (NIH)
Record Dates: First submitted 2025-03-24; First posted 2025-04-04 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Depression in Old Age
Keywords: Elder neglect; Self neglect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- APS Treatment as Usual (Active Comparator)
  Interventions: Behavioral: APS Treatment as Usual
- Intervention-Behavioral Activation (BA) (Experimental)
  Interventions: Behavioral: Intervention-Behavioral Activation (BA)

INTERVENTIONS:
Behavioral: APS Treatment as Usual — APS agencies conduct in-home investigations of alleged abuse and neglect against disabled and older adults. Investigations result in short-term stop-gap measures, primarily brief case-management centering on referral linkage to community-based services and provision of resource allocation. No direct psychological services or treatments are provided by APS, however referral to other services is also standard.
  Arms: APS Treatment as Usual
Behavioral: Intervention-Behavioral Activation (BA) — Participants will be will be guided through 8 one-hour sessions via home telehealth by the study community health worker. Each weekly < 60 minute BA session will include modules focusing on 1) Psychoeducation for depression and techniques for self-management, including pharmacologic and psychosocial treatment options; 2) Introduction of BA and guided problem-solving techniques to enhance self efficacy for managing depression and other chronic illnesses; 3) BA and problem-solving techniques to support medication management and adherence strategies; 4) BA to develop strategies and techniques for communicating with health providers and/or support resources to foster positive mood and self management; and 5) Developing a relapse prevention plan, which includes identifying triggers for lower functioning, support resources, and practice of BA techniques.
  Arms: Intervention-Behavioral Activation (BA)

SUMMARY:
The purpose of this study is to test the feasibility and acceptability of an evidence-based treatment for depression delivered over an ipad, computer, or smartphone can help Adult Protective Services (APS) clients with their activities of daily living to evaluate whether reductions on measures of depression and apathy (a) mediate reduced Elder Neglect/Self Neglect (EN/SN) behaviors; and (b) whether secondary posited mediating mechanisms are also active in impacting depression and apathy

ELIGIBILITY:
Inclusion Criteria:

* APS Case in APS Region VI- Must have open case
* PHQ 9 score- Must have score of nine (9) or more

Exclusion Criteria:

* Previous mental health diagnosis of bipolar disorder, psychotic disorders, and moderate to severe dementia
* Assessment of Consent Proxy- Those who need assessment of consent proxy
* Suicidal Intent (as indexed by PhQ-9 question 9)- Those scoring 2 or 3
* Current Alcohol and Drug Dependency- As evidenced by Cut down, Annoyed, Guilty, and Eye-opener (CAGE) score of 3 or more

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-21 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in depression as assessed by the Patient Depression Questionnaire (PHQ-9) | baseline, post-treatment ( 8 weeks after baseline), and 3 months
  This is 9 item questionnaire and each is scored from 0 (not at all) to 3 (nearly every day), for a maximum score of 27, higher score indicating more depression
Change in apathy as assessed by the Apathy Motivations Index (AMI) | baseline, post-treatment ( 8 weeks after baseline), and 3 months
  This is an 18 item questionnaire and each item is scored on a scale from 0(completely true) to 4(completely untrue), for a maximum score of 72, with higher scores indicating greater apathy
Change in Elder Neglect/Self Neglect (EN/SN) as evidenced by study developed goal attainment scale | baseline, post-treatment ( 8 weeks after baseline), and 3 months
  Participants will be given a list of 19 common daily activities and will be asked to pick one or more activities form the list that they would like to start doing or do more regularly each day or week.Each activity will be then scored based on the following scoring criteria, higher score indicating better outcome :
  (Much less than expected)-2 (Somewhat less than expected)-1 (Expected client outcome)0 (Somewhat better than expected)+1 (Much better than expected)+2

SECONDARY OUTCOMES:
Change in social connection as assessed by the Lubben Social Network Scale | baseline, post-treatment ( 8 weeks after baseline), and 3 months
  This is a 6 item questionnaire and each is scored from 0(none) to 5(none or more contacts) for a total score range of 0-30 higher scores indicating better outcome
Change in social isolation as assessed by Patient-Reported Outcomes Measurement Information System (PROMIS 8) | baseline, post-treatment ( 8 weeks after baseline), and 3 months
  This is an 8 item questionnaire and each is cored from 1(never) -5 (always) for a maximum score of 40, higher score indicating worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Leila Wood, PhD, MSSW, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No